CLINICAL TRIAL: NCT04617574
Title: A Randomized Study Comparing Endostaplers in Sleeve Gastrectomy
Brief Title: Endostapler Sleeve Gastrectomy Study
Status: Completed | Type: Observational
Sponsor: Lexington Medical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Endostapler02
Record Dates: First submitted 2020-11-02; First posted 2020-11-05 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- AEON Endostapler: Stapling performed with AEON Endostapler
  Interventions: Device: AEON Endostapler
- Endo GIA Reloads with Tri-Staple Technology: Stapling performed with Endo GIA Reloads with Tri-Staple Technology
  Interventions: Device: Endo GIA Reloads with Tri-Staple Technology

INTERVENTIONS:
Device: AEON Endostapler — Surgery with AEON Endostapler
  Groups: AEON Endostapler
Device: Endo GIA Reloads with Tri-Staple Technology — Surgery with Endo GIA Reloads with Tri-Staple Technology
  Groups: Endo GIA Reloads with Tri-Staple Technology

SUMMARY:
The goal of this prospective, post-market study is to measure AEON™ Endostapler performance for laparoscopic sleeve gastrectomy surgery versus the Endo GIA™ Reloads with Tri-Staple™ Technology from Medtronic.

DETAILED DESCRIPTION:
Stapler performance will be evaluated primarily by incidence and degree of staple line bleeding from endoscopic images, evaluated by a blinded third-party. The study will include 60 total consecutive cases of individuals undergoing a planned laparoscopic sleeve gastrectomy (LSG). The LSG procedure will be performed according to institutional standard-of-care and all subjects will undergo standard preoperative evaluation as well as post-operative care.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing planned laparoscopic sleeve gastrectomy
* Informed consent for study obtained and signed from each subject

Exclusion Criteria:

* Planned open surgical approach
* Use of staple line reinforcement material (buttress)
* Revision or other bariatric procedure
* Patients with a bleeding disorder: known coagulopathy, or Platelets <100,000, or Partial Thromboplastin Time (PTT) >45sec, or Prothrombin Time (PT) >15sec, or International Normalized Ratio (INR) >1.5
* Patients with active HIV or Hepatitis B
* Patients under the age of 18 on the date of the surgery
* Patients who are pregnant
* Patients using tobacco products within the last 2 weeks prior to surgery date
* Patients using cortisone or related products within the last 2 weeks prior to surgery date

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 subjects
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Holyoke Medical Center, Holyoke, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AEON Endostapler | Endo GIA Reloads With Tri-Staple Technology
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AEON Endostapler | Endo GIA Reloads With Tri-Staple Technology | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (16.0) | 42.8 (11.1) | 43.0 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 52
  Male | 5 | 3 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 39.5 (5.4) | 39.4 (5.3) | 39.5 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Endoscopic Staple Line Bleeding Score
Description: Intraoperative staple line bleeding score from endoscopic images as measured by the provided Bleeding Severity Scale (1 = No bleeding; 2 = Minimal bleeding; 3= Moderate bleeding; 4 = Excessive bleeding; 5 = Profuse bleeding). A lower value represents a better outcome.
Time Frame: Within surgery, after the last stapler firing
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AEON Endostapler | Endo GIA Reloads With Tri-Staple Technology
Number analyzed (Participants) | 30 | 30
score on a scale | 1.63 (.57) | 2.00 (.55)

2. Primary Outcome: Intraoperative Laparoscopic Staple Line Bleeding Score
Description: Intraoperative staple line bleeding score from laparoscopic images as measured by the provided Bleeding Severity Scale (1 = No bleeding; 2 = Minimal bleeding; 3= Moderate bleeding; 4 = Excessive bleeding; 5 = Profuse bleeding). A lower value represents a better outcome.
Time Frame: Within surgery, images captured 10 seconds after the last stapler firing
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AEON Endostapler | Endo GIA Reloads With Tri-Staple Technology
Number analyzed (Participants) | 30 | 30
score on a scale | 1.55 (.67) | 1.98 (.74)

3. Secondary Outcome: Number of Participants With Postoperative Leakage Requiring Intervention
Description: Number of participants with postoperative leakage requiring intervention
Time Frame: Within 30-day post-operative period
Measure: Count of Participants; unit: Participants
Arm/Group | AEON Endostapler | Endo GIA Reloads With Tri-Staple Technology
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Intraoperative or Postoperative Blood Transfusion
Description: Number of participants with intraoperative or postoperative blood transfusion
Time Frame: Within 72 hours of surgery start time
Measure: Count of Participants; unit: Participants
Arm/Group | AEON Endostapler | Endo GIA Reloads With Tri-Staple Technology
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Reported Device-related Adverse Events
Description: Number of participants with reported device-related adverse events
Time Frame: Within 30-day post-operative period
Measure: Count of Participants; unit: Participants
Arm/Group | AEON Endostapler | Endo GIA Reloads With Tri-Staple Technology
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Product Malfunction
Description: Number of participants with product malfunction. Product malfunction means any occurrence during the surgery where the stapler does not perform as intended.
Time Frame: Within surgery
Measure: Count of Participants; unit: Participants
Arm/Group | AEON Endostapler | Endo GIA Reloads With Tri-Staple Technology
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | AEON Endostapler | Endo GIA Reloads With Tri-Staple Technology
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT04617574/Prot_SAP_000.pdf